CLINICAL TRIAL: NCT02026232
Title: Metabolic Effects of Hydroxychloroquine
Acronym: MetaHcQ
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 & loss of funding
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 201110258; 201110258 (Other: Washington University)
Record Dates: First submitted 2013-12-24; First posted 2014-01-01 (Estimated); Results first posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes; Overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- hydroxychloroquine (Active Comparator): hydroxychloroquine twice daily for 4 weeks
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): hydroxychloroquine placebo twice daily for 4 weeks
  Interventions: Other: Hydroxychloroquine Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — 200mg twice daily
  Other Names: Plaquenil; Quineprox
  Arms: hydroxychloroquine
Other: Hydroxychloroquine Placebo — 200mg placebo twice daily
  Other Names: placebo
  Arms: Placebo

SUMMARY:
The basic plan of the study is to randomize otherwise healthy subjects with type 2 diabetes to hydroxychloroquine, 200 mg twice daily or placebo.

DETAILED DESCRIPTION:
Hydroxychloroquine is a medicine that has been used for a long time to treat patients with malaria, rheumatoid arthritis, lupus and other conditions. It is closely related to chloroquine but with a better side effect profile for long term use. In treating these conditions it was discovered to have some beneficial properties like lowering cholesterol and lowering sugar in the blood of those who have diabetes. The mechanisms underlying these effects are unknown. In animal studies, we have discovered that chloroquine appears to decrease glucose, lower blood pressure and decrease atherosclerosis (hardening of the arteries). This collection of problems commonly occurs in the metabolic syndrome and diabetes mellitus, which affects over 20% and 7% of adults in Western countries respectively. We have recently looked at the effects of chloroquine on the metabolic syndrome in humans which showed that small doses given for a short period of time would reduce insulin resistance in patients with the metabolic syndrome. Several population studies have shown similar effects with hydroxychloroquine. Since hydroxychloroquine is similar to chloroquine, we thus expect similar effects on blood glucose, blood pressure and blood cholesterol in type 2 diabetes. This offers a unique opportunity to develop a novel approach for lowering blood pressure, lipids (cholesterol and triglycerides), and glucose in people at risk for heart disease

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the age of 18 and 75, either gender, any ethnic group
* Subjects must have type 2 diabetes and the following:
* A1c of 6.5-9.0%
* Treated with at least 1000 mg of metformin daily with or without a dipeptidyl peptidase-4(DPP4)inhibitor, a sulfonylurea (glipizide, glyburide, glimepiride),bromocriptine or colesevelam.
* Subjects should have a BMI >27

Exclusion Criteria:

* Prior treatment with chloroquine or hydroxychloroquine as follows:

  1. any exposure in the past 2 years,
  2. >30 days of therapy if exposure was between 2 and 5 years ago,
  3. >90 days of therapy if exposure was between 5 and 10 years ago,
  4. >6 months of therapy if exposure was 10 to 20 years ago,
  5. >1 year of therapy if exposure was 20 to 30 years ago,
  6. No limit if last exposure was >30 years ago, e.g. during the Vietnam conflict.
* Morbid obesity (BMI >45)
* Coronary artery disease or other vascular disease
* History of stroke
* Serum creatinine >-4 mg/dl for women and >-5 mg/dl for men.
* Seizure disorder
* History of psoriasis
* Hematologic disorders, including anemia (WHO criteria for anemia:hemoglobin <13g/dL in men and <12 g/dL in women)
* Current malignancy or active treatment for recurrence prevention,e.g. tamoxifen. Cancer considered to be cured, either as a result of surgery or other treatment is not exclusionary.
* Asthma requiring daily beta agonist therapy or intermittent oral steroids is exclusionary. Inhaled steroids are acceptable. Obstructive sleep apnea will be allowed if continuous positive airway pressure(CPAP) or other therapy has been stable for 6 months. Other active respiratory diseases are excluded.
* Treatment with 50mg or greater of Metoprolol or treatment with digoxin
* Liver disease, or Liver Function Test >2 times normal
* Active infection (including HIV)
* Serious illness requiring ongoing medical care or medication
* Treatment with atypical anti-psychotic medication. Treatment with any other medication for psychiatric illness, unless on a stable dose for 6 weeks prior to enrollment. Patients with unstable psychiatric disorders are excluded per the decision of the study MD regardless of medication history.
* Taking any of the following lipid lowering medications: niacin, fibrates, and greater than 1 gm/day of fish oils
* Uncontrolled hypertension (BP >150/90 mm Hg) at enrollment
* Need for daily Over The Counter medications, or currently taking cimetidine or >1000 IU vitamin E daily and unwilling to reduce or discontinue vitamin E or discontinue cimetidine for the duration of the study. Patients taking more than 1000 IU vitamin E daily should reduce or discontinue the vitamin for 30 days before randomization.
* Pregnant or lactating women, or women intending to become pregnant
* Women not using adequate birth control (hormonal birth control is acceptable, also double barrier)
* QT corrected >450 msec on screening ECG
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-03; Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clay F. Semenkovich, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rao Kondapally Seshasai S, Kaptoge S, Thompson A, Di Angelantonio E, Gao P, Sarwar N, Whincup PH, Mukamal KJ, Gillum RF, Holme I, Njolstad I, Fletcher A, Nilsson P, Lewington S, Collins R, Gudnason V, Thompson SG, Sattar N, Selvin E, Hu FB, Danesh J; Emerging Risk Factors Collaboration. Diabetes mellitus, fasting glucose, and risk of cause-specific death. N Engl J Med. 2011 Mar 3;364(9):829-841. doi: 10.1056/NEJMoa1008862. PMID 21366474
- [Background] Schramm TK, Gislason GH, Kober L, Rasmussen S, Rasmussen JN, Abildstrom SZ, Hansen ML, Folke F, Buch P, Madsen M, Vaag A, Torp-Pedersen C. Diabetes patients requiring glucose-lowering therapy and nondiabetics with a prior myocardial infarction carry the same cardiovascular risk: a population study of 3.3 million people. Circulation. 2008 Apr 15;117(15):1945-54. doi: 10.1161/CIRCULATIONAHA.107.720847. Epub 2008 Mar 31. PMID 18378618
- [Background] Schneider JG, Finck BN, Ren J, Standley KN, Takagi M, Maclean KH, Bernal-Mizrachi C, Muslin AJ, Kastan MB, Semenkovich CF. ATM-dependent suppression of stress signaling reduces vascular disease in metabolic syndrome. Cell Metab. 2006 Nov;4(5):377-89. doi: 10.1016/j.cmet.2006.10.002. PMID 17084711
- [Background] Marmor MF, Kellner U, Lai TY, Lyons JS, Mieler WF; American Academy of Ophthalmology. Revised recommendations on screening for chloroquine and hydroxychloroquine retinopathy. Ophthalmology. 2011 Feb;118(2):415-22. doi: 10.1016/j.ophtha.2010.11.017. PMID 21292109
- [Background] Su Y, Swift M. Mortality rates among carriers of ataxia-telangiectasia mutant alleles. Ann Intern Med. 2000 Nov 21;133(10):770-8. doi: 10.7326/0003-4819-133-10-200011210-00009. PMID 11085839
- [Background] Razani B, Feng C, Semenkovich CF. p53 is required for chloroquine-induced atheroprotection but not insulin sensitization. J Lipid Res. 2010 Jul;51(7):1738-46. doi: 10.1194/jlr.M003681. Epub 2010 Mar 5. PMID 20208057
- See also: Washington University Research Patient Registry — https://rpr.wustl.edu/
- See also: Clay F. Semenkovich, M.D. — http://endo.wustl.edu/clay-f-semenkovich-m-d/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants withdrew consent prior to the baseline visit. After the baseline visit, participants were randomized to either the hydroxychloroquine group or the placebo group.
Period: Overall Study
Arm/Group | Hydroxychloroquine | Placebo
Started | 10 | 11
Completed | 7 | 9
Not Completed | 3 | 2
Not completed — incomplete visit/missing data | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine | Placebo | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (14) | 61 (7) | 59 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 3 | 8 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5 | 8 | 13
  African American | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Effect of HCQ on Fasting Blood Glucose
Description: determined by fasting blood glucose performed at baseline and follow-up
Time Frame: 4 weeks
Population: randomized participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 7 | 9
mg/dL
  Baseline Glucose (mg/dL) | 186.9 (64.5) | 163.1 (22.5)
  Follow-up Glucose (mg/dL) | 165.9 (67.1) | 158.8 (38.7)
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.05, t-test, 2 sided

2. Secondary Outcome: Effect of HCQ on Fasting Low Density Lipoprotein
Description: determined by lipid profile with calculated LDL performed at baseline and follow-up
Time Frame: 4 weeks
Population: Randomized Participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 7 | 9
mg/dL
  Baseline - LDL (mg/dL) | 90.4 (21.4) | 92.8 (26.2)
  Follow-up - LDL (mg/dL) | 72.4 (21.6) | 87.7 (23.8)

ADVERSE EVENTS:
Time Frame: Adverse events will be monitored during the study -- approximately 1 month of study participation
Arm/Group | Hydroxychloroquine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 3/10 | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=10) | Placebo (N=11)
Drop in hematocrit (Blood and lymphatic system disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-05-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT02026232/Prot_SAP_000.pdf